CLINICAL TRIAL: NCT05469724
Title: Clinical Characteristics and Outcome Registry in Patients Admitted With Acute Pulmonary Embolism
Brief Title: Clinical Pulmonary Embolism
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Peter Samir Roshdy, Clinical characteristics of acute pulmonary embolism, Assiut University
Other Study IDs: Clinical of acute pulm emb
Record Dates: First submitted 2022-06-01; First posted 2022-07-22 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-04

CONDITIONS: Acute Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Role of ct pulmonary angiography in diagnosis of pulmonary embolism — Role of ct pulmonary angiography in diagnosis of acute pulmonary embolism as filling defect in pulmonary artery

SUMMARY:
To evaluate the clinical characteristics, risk factors, management and outcome of patients admitted e acute pulmonary embolism in chest diseases department and Respiratory Icu in Assiut University hospital

DETAILED DESCRIPTION:
Pulmonary embolism (PE) occurs when there is a disruption to the flow of blood in the pulmonary artery or its branches by a thrombus that originated somewhere else. In deep vein thrombosis (DVT), a thrombus develops within the deep veins, most commonly in the lower extremities. PE usually occurs when a part of this thrombus breaks off and enters the pulmonary circulation. Very rarely, PE can occur from the embolization of other materials into the pulmonary circulation such as air, fat, or tumor cells.Risk factors can be classified as genetic and acquired. Genetic risk factors include thrombophilia such as factor V Leiden mutation, prothrombin gene mutation, protein C deficiency, protein S deficiency, hyperhomocysteinemia, among others. Acquired risk factors include immobilization for prolonged periods (bed rest greater than three days, anyone traveling greater than 4 hours, whether by air, car, bus, or train), recent orthopedic surgery, malignancy, indwelling venous catheter, obesity, pregnancy, cigarette smoking, oral contraceptive pill use

Other predisposing factors for VTE include:

Fracture of lower limb Hospitalization for heart failure or atrial fibrillation/flutter within the previous three months Hip or knee replacement Major trauma History of previous venous thromboembolism Central venous lines Chemotherapy Congestive heart failure or respiratory failure Hormone replacement therapy Oral contraceptive therapy Postpartum period Infection (specifically pneumonia, urinary tract infection, and HIV) Cancer (highest risk in metastatic disease) Thrombophilia Bed rest greater than three days Obesity Pregnancy Cancer carries a high risk for thrombus formation and hence, PE. Pancreatic cancer, hematological malignancies, lung cancer, gastric cancer, and brain cancer carry the highest risk for VTThe most common symptoms of PE include the following: dyspnea, pleuritic chest pain, cough, hemoptysis, presyncope, or syncope. Dyspnea may be acute and severe in central PE, whereas it is often mild and transient in small peripheral PE. In patients with preexisting heart failure or pulmonary disease, worsening dyspnea may be the only symptom. Chest pain is a frequent symptom and is usually caused by pleural irritation due to distal emboli causing pulmonary infarction.

ELIGIBILITY:
Inclusion Criteria:

* Patients above 18 years old and less than 75 year old

Exclusion Criteria:

* patients with chronic thromboembolism _patient less than 18 years old

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study of patient between 18and 75 year presented by acute pulmonary embolism
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-07 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
European society of cardiology risk score and its measurement units | 1 year
  Classification of patients admitted with acute pulmonary embolism into high risk ,low risk, intermediate high and intermediate low risk

SECONDARY OUTCOMES:
Pulmonary embolism severity index risk score and its units of measurement | 1 year
  Classification of patients according to rik score of pulmonary embolism severity index

REFERENCES:
- [Background] Howard L. Acute pulmonary embolism. Clin Med (Lond). 2019 May;19(3):243-247. doi: 10.7861/clinmedicine.19-3-247. PMID 31092519
- [Background] Hepburn-Brown M, Darvall J, Hammerschlag G. Acute pulmonary embolism: a concise review of diagnosis and management. Intern Med J. 2019 Jan;49(1):15-27. doi: 10.1111/imj.14145. PMID 30324770
- [Background] Rivera-Lebron B, McDaniel M, Ahrar K, Alrifai A, Dudzinski DM, Fanola C, Blais D, Janicke D, Melamed R, Mohrien K, Rozycki E, Ross CB, Klein AJ, Rali P, Teman NR, Yarboro L, Ichinose E, Sharma AM, Bartos JA, Elder M, Keeling B, Palevsky H, Naydenov S, Sen P, Amoroso N, Rodriguez-Lopez JM, Davis GA, Rosovsky R, Rosenfield K, Kabrhel C, Horowitz J, Giri JS, Tapson V, Channick R; PERT Consortium. Diagnosis, Treatment and Follow Up of Acute Pulmonary Embolism: Consensus Practice from the PERT Consortium. Clin Appl Thromb Hemost. 2019 Jan-Dec;25:1076029619853037. doi: 10.1177/1076029619853037. PMID 31185730
- [Background] Righini M, Robert-Ebadi H. Diagnosis of acute Pulmonary Embolism. Hamostaseologie. 2018 Feb;38(1):11-21. doi: 10.5482/HAMO-17-07-0023. Epub 2018 Feb 26. PMID 29536476
- [Background] Sin D, McLennan G, Rengier F, Haddadin I, Heresi GA, Bartholomew JR, Fink MA, Thompson D, Partovi S. Acute pulmonary embolism multimodality imaging prior to endovascular therapy. Int J Cardiovasc Imaging. 2021 Jan;37(1):343-358. doi: 10.1007/s10554-020-01980-9. Epub 2020 Aug 30. PMID 32862293
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/31588070/